CLINICAL TRIAL: NCT01692431
Title: The Impact of Fish-oil Fatty Acids on Postprandial Vascular Reactivity
Acronym: FOFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12/EE/011
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Physiological Phenomena; Endothelial Nitric Oxide Synthase; Eicosapentaenoic Acid; Docosahexaenoic Acid (All-Z Isomer)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DHA (Experimental): High fat meal containing DHA rich oil.
  Interventions: Dietary Supplement: DHA
- EPA (Experimental): High fat meal containing EPA.
  Interventions: Dietary Supplement: EPA
- Control (Placebo Comparator): High fat meal with no/negligable omega-3 fatty acid content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA — High fat meal containing EPA
  Arms: EPA
Dietary Supplement: DHA — High fat meal containing DHA
  Arms: DHA
Dietary Supplement: Placebo — High fat meal containing negligible EPA/DHA content
  Arms: Control

SUMMARY:
The primary aim of this study is to determine the impact of individual fish oil fatty acids on vascular reactivity and to identify underlying physiological and molecular mechanism of any observed effects. In addition response to intervention according to genotype will be determined retrospectively.

DETAILED DESCRIPTION:
A loss of vascular reactivity and increased vascular tone is being increasingly recognised as a significant cardiovascular disease (CVD) risk factor and highly predictive of future CVD events. A previous study by our group has shown the inclusion of a fish oil mixture administered alongside a high fat meal preserves postprandial vascular function in healthy men [1]. In this three arm, placebo controlled cross over study, the impact of individual fatty acids contained within fish-oil on postprandial vascular reactivity (measured at 4 hour post test meal) will be assessed for the first time. Clinical measurements of vascular function which correlate with CVD risk factors and are predictive of future CVD events will be undertaken in order to assess any potentially beneficial effects. In addition plasma samples will be taken at 0 and 4 hours to determine the change in concentration of modulators of vascular tone. Accordingly, our nutrients of interest which will be administered in the intervention arms of the study, will be present in this lipoprotein rich fraction. By exposing cells in culture to these EPA- and DHA-enriched lipoproteins, mechanisms underlying the vascular response in our human volunteers will be investigated. Finally we will measure the plasma fatty acid profile to confirm that circulating concentrations of EPA and DHA are increasing postprandially according to intake.

As it is now recognised that genetic variation, in addition to being an important determinant of the risk of all known chronic diseases, plays a large part in determining an individual's response to dietary change, DNA will be extracted from whole blood taken at the clinical screening and stored for subsequent genotyping for variants likely to be important in the regulation of EPA and DHA metabolism and vascular tone. Although the current study will not be fully powered to generate definite conclusion regarding genotype*diet interactions, it will serve to generate pilot data for future studies.

ELIGIBILITY:
Inclusion Criteria:

In order to recruit a population at a relative risk of developing CVD of >1.5 males aged 35-55 years, who possess one of the following risk factors for CVD will be recruited through local advertisement:

* Total cholesterol > 6mmol/L
* High density lipoprotein cholesterol (HDLC) < 1.0mmol/L
* Systolic blood pressure > 140 mmHg
* Diastolic blood pressure > 90 mmHg
* Waist circumference > 102cm

Exclusion Criteria:

Current smokers, or ex-smokers ceasing < 3 months ago

Subjects with existing or significant past medical history of vascular disease or any medical condition likely to affect the study measures e.g. vascular disease, circulatory (i.e. Reynaud's), diabetes, systemic lupus erythematosus, hepatic, renal, digestive, haematological, neurological, cancer or thyroidal disease.

Those with known allergies to the intervention foods / commercially available supplements.

Those unprepared to adhere to dietary restrictions during the trial i.e. for 3 days preceding each assessment visit (and for a 3 day run-in period) or unwilling to comply with the assessments per protocol.

Parallel participation in another research project which involves concurrent dietary intervention and/or sampling of biological fluids/material.

Having vaccinations (excluding the flu vaccination) or antibiotics within 3 months of start of trial, and those with vaccinations scheduled for during the trial.

Taking EPA or DHA containing food / dietary supplements likely to affect the study results e.g. supplements derived from marine organisms which equate to a greater than 1 gram of EPA and DHA per daily serving. Prospective participants who are willing to cease supplementation 2 month preceding, and during, the trial will be considered on a case by case basis.

Habitual consumption of more than one portion of oily fish per week (as defined as 140g of any oil fish, including salmon, trout, mackerel, sardines, pilchards, herring, kipper, eel, whitebait, etc).

Prescribed lipid lowering, medicine affecting lipoprotein metabolism or blood blotting, hypertension, vasodilators (e.g. Viagra) or antibiotic medication.

Assessed from the clinical screening.

Unsatisfactory biochemical or haematological assessment assessed by the studies clinical advisor

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Endopat | Change from baseline at 4 hours postprandially
  EndoPat is an easy to use and rapid technique which has been validated against other clinically accepted measures of endothelial function such as Flow Mediated Dilation and Coronary Blood Flow measured by angiography alongside acetylcholine infusion. EndoPat has also been shown to correlate with multiple known CVD risk factors and to be predictive of future cardiovascular events. In addition, EndoPat will be utilised alongside oral administration of nitroglycerin in order to establish if peripheral arterial tone is altered in response to EPA or DHA in a non-Nitric Oxide dependent manner. EndoPAT produces a reactive hyperaemic index score which is indicative of the endothelial's capacity to produce NO, which itself is indicative of general endothelial function. EndoPAT will be assessed using a standardised methodology developed by Itamar Medical, which involves measuring changes in dilation in response to induced hyperaemia.

SECONDARY OUTCOMES:
Pulse Wave Velocity | Change from baseline at 4 hours postprandially
  Pulse Wave Velocity (PWV) analysis will also be utilised in order to measure arterial stiffness. PWV analysis will allow several non-invasive measurements to be taken simultaneously including PWV, which is an established index of arterial stiffness, and augmentation index, an indirect measure of arterial stiffness which is dependent on wave-reflections and independent of pulse pressure. PWV and associated measures will be measured using methodology developed by Skidmore medical. PWV is measured in m/sec while augmentation index is measured as a % of augmentation (of central aortic pressure by a reflected pulse wave).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Minihane, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Norwich Medical School, Norwich, United Kingdom

REFERENCES:
- [Background] Armah CK, Jackson KG, Doman I, James L, Cheghani F, Minihane AM. Fish oil fatty acids improve postprandial vascular reactivity in healthy men. Clin Sci (Lond). 2008 Jun;114(11):679-86. doi: 10.1042/CS20070277. PMID 18052925